CLINICAL TRIAL: NCT02938156
Title: Evaluation of Real World Outcomes With Extended Half-Life Concentrates for Routine Clinical Use in Haemophilia A and B: UK - EHL Outcomes Registry
Brief Title: UK - EHL Outcomes Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Pratima Chowdary, Consultant Haematologist, Royal Free Hospital NHS Foundation Trust
Other Study IDs: RFH/9782
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe haemophilia A and B (SHA, SHB) are inherited bleeding disorders affecting male patients and are characterised by low levels of circulating clotting factors VIII and IX respectively. Clinically low levels present with multiple recurrent bleeds into joints and muscle from the first couple of years of life. In addition patients may present with spontaneous and potentially fatal bleeding into any organ. The mainstay of treatment is replacement with the missing factor in the form of intravenous injections of factor VIII and IX. Clotting factors can be given to treat a bleed or can be given to prevent a bleed, and the latter is termed prophylaxis. Regular prophylaxis is the current standard of care and aims to decrease spontaneous bleeding events and resulting joint damage, and this requires patients to self-infuse factor into their veins two to four times week. Patient's compliance with prescribed regimen and recommendations has a significant influence on outcomes.

Advances in biomolecular and protein engineering have extended the duration of the effect of clotting factor VIII and IX through multiple mechanisms. This extension of the duration of the effect presents the clinician and patients with opportunities to tailor the treatment to their particular needs, circumstances and body other characteristics. It has been suggested that decreasing the frequency of infusions will improve adherence and thus contribute to improved outcomes.

In rare disorders, it is an accepted fact that post-marketing studies are crucial to understand the generalisability of the efficacy and safety outcomes and identify any new safety and efficacy concerns in relation to specific population group. The investigators propose the development of a registry for systematic collection of information with the dual aim of analysing the relationship between patient and treatment characteristics, and outcomes, and simultaneously identify areas for practice development that can improve the overall quality of life experienced by the haemophilia patient community.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Haemophilia A or B requiring replacement therapy
2. Patients or parents able to provide informed consent
3. Patients being considered for use of EHL - CFC.

Exclusion Criteria:

1. Patients currently enrolled into a clinical trial of investigational medicinal product.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Haemophilia A or B requiring replacement therapy or being considered for use of EHL - CFC.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12-17 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Bleed Control | 2 years post enrolment
  Investigate changes to bleed control using questionnaire & Haemtrack (software package to record therapy received
Joint Health | 2 years post enrolment
  Target joint assessment and questionnaire

SECONDARY OUTCOMES:
EQ-5D-5L | 2 years post enrolment
  Patient Questionnaire
HAEM-A-QoL | 2 years post enrolment
  Patient Questionnaire
Haemo-QoL | 2 years post enrolment
  Patient Questionnaire
Physical Activity QoL | 2 years post enrolment
  Patient Questionnaire
Haemoprefer | 2 years post enrolment
  Patient Questionnaire
Identify the value of individualised prophylaxis | 5 years
  Patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, Principal Investigator — Royal Free Hospitals NHS Foundation Trust
Locations (21):
- United Kingdom (21):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Birmingham Women and Childrens, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital Bristol, Bristol
  - Kent & Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - University of Coventry & Warwickshire, Coventry
  - Glasgow Royal Hospital for Children, Glasgow
  - Royal Infirmary, Glasgow
  - Lincoln County Hospital, Lincoln
  - Liverpool University Hospital, Liverpool
  - Royal Free Hospital NHS Foundation Trust, London
  - Great Ormond Street Hospital, London
  - Hammersmith Hospital, London
  - St George's Hospital, London
  - Royal Victoria Hospital, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - Churchill Hospital Oxford, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - Sheffield Children's Hospital, Sheffield
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Koopman SF, Goedhart TMHJ, Bukkems LH, Mulders TM, Leebeek FWG, Fijnvandraat K, Coppens M, Mathias M, Collins PW, Tait RC, Bagot CN, Curry N, Payne J, Chowdary P, Cnossen MH, Mathot RAA; OPTI-CLOT study group and SYMPHONY consortium. A new population pharmacokinetic model for recombinant factor IX-Fc fusion concentrate including young children with haemophilia B. Br J Clin Pharmacol. 2024 Jan;90(1):220-231. doi: 10.1111/bcp.15881. Epub 2023 Sep 12. PMID 37567779